CLINICAL TRIAL: NCT00114049
Title: A Pivotal Phase III, Single Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Dose-Ranging Study to Investigate the Efficacy and Safety of Single Oral Doses of 10mg, 25mg, 50mg and 70mg GW406381 and 550mg Naproxen Sodium in Subjects With Pain Following Third Molar Tooth Extraction
Brief Title: Dental Pain (Following Third Molar Tooth Extraction) Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CXA30001
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Dental Pain; Surgery, Dental
Keywords: Dental Pain; Dental Surgery; Cox-2 inhibitor
MeSH Terms: conditions — Toothache | interventions — GW406381X

INTERVENTIONS:
Drug: GW406381

SUMMARY:
The purpose of this study is to evaluate the effectiveness of GW406381 (a COX-2 inhibitor) in treating the signs and symptoms of dental pain following third molar tooth extraction.

DETAILED DESCRIPTION:
A Pivotal Phase III, Single Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Dose-Ranging Study to Investigate the Efficacy and Safety of Single Oral Doses of 10mg, 25mg, 50mg, and 70mg GW406381 and 550mg Naproxen Sodium in Subjects With Pain Following Third Molar Tooth Extraction

ELIGIBILITY:
Inclusion criteria:

* Scheduled for outpatient surgical removal of at least two third molar teeth.

Exclusion criteria:

* Subjects who do not achieve moderate to severe pain.
* Subjects who do not use acceptable contraception.
* Additional medical criteria will be assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-12; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Difference between treatments over time based on pain intensity and pain relief scores.

SECONDARY OUTCOMES:
Difference between treatments based on changes in onset, duration of activity, overall effectiveness, and patient based assessments.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States